CLINICAL TRIAL: NCT03968445
Title: Neuroinflammation After Myocardial Infarction - Imaging Substudy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, M.D. P.h.D., Director for the Division Molecular Imaging and Therapeutics, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-300003221 R19-045
Record Dates: First submitted 2019-05-16; First posted 2019-05-30 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Recent Myocardial Infarction (Experimental)
  Interventions: Drug: [18F]DPA-714-PET/MRI
- undergoing elective percutaneous coronary intervention (Experimental)
  Interventions: Drug: [18F]DPA-714-PET/MRI

INTERVENTIONS:
Drug: [18F]DPA-714-PET/MRI — [18F]DPA-714-PET/MRI

SUMMARY:
The purpose of the study is to see if positron emission tomography and magnetic resonance imaging (PET/MRI) with an investigational drug called [18F]DPA-714 will show inflammation in the brain after a heart attack. This study may help physicians and researchers better understand the role of brain inflammation in heart disease and develop new treatments to protect the brain.

DETAILED DESCRIPTION:
The primary objective of this study is to measure the concentration and the regional brain distribution of activated brain microglia/macrophages using the PET ligand [18F]DPA-714 in individuals with recent AMI. The basic premise is that AMI leads to systemic inflammation that includes inflammation in the brain. The PET tracer [18F]DPA-714 binds to the 18 kDa translocator protein (TSPO, also known as the peripheral benzodiazepine receptor) in the mitochondria of activated microglia/macrophages and provides a non-invasive measure of neuroinflammation. The estimates of brain TSPO binding in patients with recent AMI will be compared to a matched group of patients who have undergone a recent elective PCI procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in UAB IRB protocol "Neuroinflammation After Acute Myocardial Infarction" (IRB-300002751, PI Lazar).
2. 21 years of age or older
3. . English speaking with at least 8th grade education
4. High or mixed affinity binder for TSPO ligands based on genotyping for single nucleotide polymorphism (SNP) rs6971.
5. Admission to UAB Hospital for ST-elevation acute myocardial infarction (AMI) and treatment with percutaneous coronary intervention (PCI) OR Undergoing elective percutaneous coronary intervention (PCI)

Exclusion Criteria:

1. Contraindication to MRI
2. Pregnancy
3. Lactation
4. Serious medical co-morbidity that may interfere with participation
5. Prior myocardial infarction
6. Severe anemia
7. Prior coronary artery bypass grafting
8. Prior angioplasty and/or coronary artery stent placement (PCI group only)
9. History of traumatic head injury defined by a loss of consciousness ≥30 minutes or seizure at the time of injury
10. Diagnosis of major depression
11. Diagnosis of dementia
12. Low affinity binder for TSPO ligands based on genotyping for SNP rs6971.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
TPSO-PET measurement of neuroinflammation after acute myocardial infarction | 2 years
  The regional brain concentrations of [F-18]DPA-714, a PET imaging marker of neuroinflammation, will be compared between study participants who have recently been hospitalized for acute myocardial infarction (AMI) and a control group undergoing elective percutaneous coronary interventions (PCI).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham Medical Center, Birmingham, Alabama, United States